CLINICAL TRIAL: NCT04214431
Title: Reducing Fear of Childbirth Among Pregnant Women: Women's Lived Experience, Predictors, and Effects of Mindfulness-based Childbirth Education
Brief Title: Reducing Fear of Childbirth Among Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N201508025
Record Dates: First submitted 2019-12-20; First posted 2020-01-02 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Fear of Childbirth
Keywords: fear of childbirth, pregnancy, childbirth education,

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Mindfulness-Based Childbirth Education (Experimental): Women in the experimental group received eight week mindfulness-based childbirth education program delivered one class each week.
  Interventions: Behavioral: Mindfulness-Based Childbirth Education
- Control group (No Intervention): Women in the control group received standardized care.

INTERVENTIONS:
Behavioral: Mindfulness-Based Childbirth Education — 8-week mindfulness-based childbirth education
  Arms: Mindfulness-Based Childbirth Education

SUMMARY:
Pregnant women often experience fear of childbirth or anxiety toward the labor pain or uncertainties associated with labor process. To develop and evaluate the efficacy of childbirth educational interventions on reduction of fear or anxiety is an important issue in maternal health care.

DETAILED DESCRIPTION:
Fear of childbirth is a common clinical problem among perinatal women and link to adverse health effects on mother's and offspring's well-being. Recently, reducing the childbirth fear becomes a highly important maternity care issues as a result of the fact that the birth rate has been declining rapidly as well as Cesarean rate increased steadily. However, the studies on fear of childbirth among perinatal population in Taiwan were limited. In this proposal the investigators plan to conduct a randomized controlled study examining the effects of mindfulness-based childbirth education. In the randomized controlled study, women will be recruited and randomized into the experiment group (receiving mindfulness-based childbirth education and traditional childbirth education),or will be allocated in the control group receiving traditional childbirth education. Intention-to-treat analysis as well as mixed regression modeling will be used to estimate the effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. aged of 20 years or greater;
2. 12-25 week of gestation, Singleton pregnancy;
3. able to communicate with Mandarin or Taiwanese;
4. High levels of fear of Childbirth (greater 9 or above on Numeric Rating Scale).

Exclusion Criteria:

1. Current having psychological diseases or substance abuse, unable to follow the mindfulness-based childbirth education;
2. unable to attend every class or each assessment;
3. received any cognitive training in past one year.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 404 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2019-02-23 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Fear of childbirth | pregnancy 12-24 weeks
  Fear of childbirth measure by the Wijma Delivery Expectancy/ Experience Questionnaires, W-DEQ with total score ranging between 0~165. The high score indicated higher levels of childbirth fear.
Fear of childbirth | pregnancy 32-36 weeks
  Fear of childbirth measure by the Wijma Delivery Expectancy/ Experience Questionnaires, W-DEQ with total score ranging 0-165. The higher score indicated higher level of childbirth fear.
Fear of childbirth | postpartum 1 week
  Fear of childbirth measure by the Wijma Delivery Expectancy/ Experience Questionnaires, W-DEQ, with total score ranging 0-165. The higher score indicated the higher level of childbirth fear.

SECONDARY OUTCOMES:
Anxiety | pregnancy 12-24 weeks
  Anxiety measure by State-Trait Anxiety Inventory, STAI
Anxiety | pregnancy 32-36 weeks
  Anxiety measure by State-Trait Anxiety Inventory, STAI, with an overall score ranging 20,80. A higher score indicates higher anxiety.
Anxiety | postpartum 1 week
  Anxiety measure by State-Trait Anxiety Inventory, STAI, with an overall score ranging 20,80. A higher score indicates higher anxiety.
Depression | pregnancy 12-24 weeks
  Depression measure by Edinburgh Postnatal Depression Scale, EPDS, , with a total score ranging 0,30. A higher score represents a higher level of depression.
Depression | pregnancy 32-36 weeks
  Depression measure by Edinburgh Postnatal Depression Scale, EPDS, , with a total score ranging 0,30. A higher score represents a higher level of depression.
Depression | postpartum 1 week
  Depression measure by Edinburgh Postnatal Depression Scale, EPDS, , with a total score ranging 0,30. A higher score represents a higher level of depression.
Mindfulness | pregnancy 12-24 weeks
  Mindfulness measure by Chinese Version Mindful Attention Awareness Scale (CMAAS), with a total score ranging 15-90, the higher score and the high levels of mindfulness.
Mindfulness | pregnancy 32-36 weeks
  Mindfulness measure by Chinese Version Mindful Attention Awareness Scale, CMAAS, with a total score ranging from 15-90, the higher score the high levels of mindfulness.
Mindfulness | postpartum 1 week
  Mindfulness measure by Chinese Version Mindful Attention Awareness Scale, CMAAS, with a total score ranging 15-90, and the higher the score, the higher levels of mindfulness.
Birth outcomes | postpartum 1 week
  To analyze the mode of delivery, including vaginal delivery or cesarean delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yu Kuo, Ph.D., Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taiwan, R.O.C., Taipei, Taiwan

REFERENCES:
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203